CLINICAL TRIAL: NCT03503864
Title: Clinical Research on Efficacy and Safety of Combined Chemotherapy With Arsenic Trioxide in Stage 4/M Neuroblastoma：A Prospective，Single-arm, Open-label, Multi-center Study
Brief Title: Phase II Study of Combined Chemotherapy With Arsenic Trioxide in Stage 4/M Neuroblastoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yang Li (Other)
Responsible Party: Sponsor-Investigator, Yang Li, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Organization: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYS-C-202007
Record Dates: First submitted 2018-01-21; First posted 2018-04-20 (Actual); Results first posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Arsenic Trioxide; Children
MeSH Terms: conditions — Neuroblastoma | interventions — Arsenic Trioxide

STUDY DESIGN:
Intervention Model Description: Combined induction chemotherapy with arsenic trioxide
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ATO-combined chemotherapy (Experimental): Patients receive combined induction chemotherapy with arsenic trioxide.
  Interventions: Drug: Arsenic Trioxide

INTERVENTIONS:
Drug: Arsenic Trioxide — Arsenic trioxide（ATO） is administered 0.16mg/kg per day over eight hours IV daily for ten days. Patients will receive ATO alone on days 1-2 and combined with conventional induction chemotherapy on days 3-10. Nine cycles at most of ATO-combined chemotherapy were applied in the whole scheme.
  Other Names: ATO

SUMMARY:
This clinical trial aims to explore and evaluate the efficacy and safety of combined chemotherapy with arsenic trioxide for stage 4/M neuroblastoma.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-lable, multi-center clinical trial. Children≤ 14 years old are eligible for this study if they were newly diagnosed with neuroblastoma and assessed as stage 4 according to the International Neuroblastoma Staging System (INSS) or stage M according to the International Neuroblastoma Risk Group (INRG) respectively. Patients enrolled in this study will receive combined induction chemotherapy with arsenic trioxide following an modifed protocol based on N7 and NB2004 protocols. Objective response rate (ORR) at 4 weeks after completing induction chemotherapy was defined as the main outcome and adverse events were monitored and graded in the meantime.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated Stage 4/M neuroblastoma patients according to the International Neuroblastoma Staging System（INSS) or the International Neuroblastoma Risk Group (INRG) staging system;
2. Patients not more than 14 years old;
3. There are measurable lesions;
4. Guardians agreed and signed informed consent.

Exclusion Criteria:

1. Patients who had suffered from other tumors and received chemotherapy or abdominal radiotherapy.
2. Patients with one or more critical organs failure such as heart, brain, kidney failure.

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2028-12-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yang Li, Professor, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Until July 31, 2023, a total of 80 children from the paediatrics departments of 8 hospitals, were recreated in this study.
Pre-assignment Details: 6 patients changed therapeutic regimen，7 patient withdrew consent.
Groups:
- ATO-combined Chemotherapy: Patients receive combined induction chemotherapy with arsenic trioxide.
  Arsenic Trioxide: Arsenic trioxide（ATO） is administered 0.18mg/kg per day over eight hours IV daily for ten days. Patients will receive ATO alone on days 1-2 and combined with conventional induction chemotherapy on days 3-10. Nine cycles at most of ATO-combined chemotherapy were applied in the whole scheme.
Period: Overall Study
Arm/Group | ATO-combined Chemotherapy
Started | 80
Completed | 67
Not Completed | 13
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 7

BASELINE CHARACTERISTICS:
Arm/Group | ATO-combined Chemotherapy
Number analyzed (Participants) | 67
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 3.5 [2.6 to 4.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 67
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  China | 67

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The percentage of patients who had complete remission（CR）or partial remission（PR）after induction chemotherapy combined ATO. Per Response Evaluation Criteria In Solid Tumors Criteria (WHO criteria) for target lesions and assessed by MRI or CT: CR: All lesions completely disappear, maintained for at least 4 weeks. PR: Estimated tumor size reduction by more than 50%, maintained for at least 4 weeks.
Time Frame: Four weeks after ATO-combined induction chemotherapy
Measure: Count of Participants; unit: Participants
Arm/Group | ATO-combined Chemotherapy
Number analyzed (Participants) | 67
Participants | 62

2. Secondary Outcome: Overall Survival Rate
Description: The proportion of patients who are alive from the date of randomization to 3 years, regardless of the cause of death.
Time Frame: 3 years.
Population: 1 patient lost to follow-up for OS.
Measure: Number (95% Confidence Interval); unit: percentage of participent
Arm/Group | ATO-combined Chemotherapy
Number analyzed (Participants) | 66
percentage of participent | 68.0 [53.8 to 78.6]

3. Secondary Outcome: Progression Free Survival Rate
Description: The proportion of patients who have not experienced progression or death from any cause, whichever occurs first, within a maximum of 3 years from the date of enrollment.
  Treatment response was evaluated according to the WHO criteria for the efficacy of solid tumours, which was classified as complete response (CR), partial response (PR), stable disease (SD) and progressive disease (PD). PD was characterized as more than 25% increase in one or more lesions or appearance of new lesions.
Time Frame: 3 years.
Population: 6 patients lost to follow-up for PFS.
Measure: Number (95% Confidence Interval); unit: percentage of participent
Arm/Group | ATO-combined Chemotherapy
Number analyzed (Participants) | 61
percentage of participent | 47.7 [32.5 to 61.4]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events are monitored and graded by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)
Time Frame: From date of ATO-combined chemotherapy until the date of first documented adverse event, and follow up for 3 years.
Measure: Count of Participants; unit: Participants
Groups:
- Myelosuppression; Vomiting; Transaminitis; Cardiovascular Toxicity; Infection: Grade 3/4 adverse events
Arm/Group | Myelosuppression | Vomiting | Transaminitis | Cardiovascular Toxicity | Infection
Number analyzed (Participants) | 67 | 67 | 67 | 67 | 67
Participants | 60 | 33 | 4 | 1 | 20

ADVERSE EVENTS:
Time Frame: Adverse Events monitored up to 3 years.
Arm/Group | ATO-combined Chemotherapy
All-Cause Mortality (participants affected / at risk) | 22/67
Serious Adverse Events (participants affected / at risk) | 0/67
Other Adverse Events (participants affected / at risk) | 67/67
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ATO-combined Chemotherapy (N=67)
Myelosuppression (Blood and lymphatic system disorders) | 67
Vomiting (Gastrointestinal disorders) | 54
Infection (Infections and infestations) | 23
Transaminitis (Hepatobiliary disorders) | 23
Cardiovascular toxicity (Cardiac disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT03503864/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/64/NCT03503864/ICF_001.pdf